CLINICAL TRIAL: NCT01941329
Title: Prospective, Randomized, Multicentre, Open-label, Phase II / III Study to Assess Efficacy and Safety of Ranibizumab 0.5 mg Intravitreal Injections Plus Panretinal Photocoagulation (PRP) Versus PRP in Monotherapy in the Treatment of Subjects With High Risk Proliferative Diabetic Retinopathy. (PROTEUS)
Brief Title: Prospective, Randomized, Multicentre, Open-label, Phase II / III Study to Assess Efficacy and Safety of Ranibizumab 0.5 mg Intravitreal Injections Plus Panretinal Photocoagulation (PRP) Versus PRP in Monotherapy in the Treatment of Subjects With High Risk Proliferative Diabetic Retinopathy.
Acronym: PROTEUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR-RET-2013-05
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: High Risk Proliferative Diabetic Retinopathy
Keywords: Diabetes; Proliferative Retinopathy; Ranibizumab; Panretinal Photocoagulation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranimizumab + Panretinal photocoagulation (PRP) (Experimental): 3 Intravitreous injections of ranibizumab combined with standard PRP (2 ± 1 weeks after injection), at month-0, month-1 and month-2 that can be repeated after month-3, with always at least 1 month of interval between injections.
  Interventions: Procedure: Panretinal Photocoagulation (PRP); Drug: Intravitreous injection of ranibizumab
- Panretinal photocoagulation (PRP) (Active Comparator): Panretinal photocoagulation treatment (PRP) between month-0 and month-2, with 1 mandatory laser session in month-0 and more laser sessions as needed until Month-2 to complete the PRP treatment.
  After completing the PRP treatment, PRP sessions can be repeated from Month-3 to Month-11.
  Interventions: Procedure: Panretinal Photocoagulation (PRP)

INTERVENTIONS:
Procedure: Panretinal Photocoagulation (PRP)
Drug: Intravitreous injection of ranibizumab
  Arms: Ranimizumab + Panretinal photocoagulation (PRP)

SUMMARY:
This study is a prospective, randomized, multicentre, open label study that intents to compare the efficacy and safety of ranibizumab 0.5 mg Intravitreal (ITV) injections plus Panretinal Photocoagulation versus Panretinal Photocoagulation alone in the regression of the neovascularization area in patients with High Risk Proliferative Diabetic Retinopathy over a 12-month treatment period.

One of the major complications of the diabetes mellitus is Diabetic Retinopathy (DR), one of the leading causes of visual impairment in working age in industrialized countries. Longer diabetes duration and poor glycaemic and blood pressure control are strongly associated with Diabetic Retinopathy. The overall prevalence of any form of Diabetic Retinopathy is 34.4% and 6.96% corresponds to Proliferative Diabetic Retinopathy (PDR). Therefore, approximately 93 million people have Diabetic Retinopathy and 17 million of them have Proliferative Diabetic Retinopathy.

It has been shown that treatment with repeated injections of ranibizumab can improve visual acuity in patients with PDR. Further, , the standard PRP treatment of PDR remains unsatisfactory. The knowledge of the mechanisms of this retinal complication is incomplete and, therefore, efforts should be done to understand and characterize patients' eyes response to combined treatments.

Therefore, the purpose of this study is to compare the standard treatment for PDR (i.e. Panretinal Photocoagulation) with Panretinal Photocoagulation treatment combined with ITV injections of ranibizumab since it is expected that anti-vascular endothelial growth factor (VEGF) treatment with ITV injections will increase the rate of success of Panretinal Photocoagulation in regression of neovascularization with improved final visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* High-risk proliferative diabetic retinopathy (HR-PDR); Neovascularization in the disc (NVD) ≥ 1/4 disc area (DA) OR Neovascularization elsewhere (NVE) ≥ 1/2 DA; NVE < 1/2 DA + vitreous and/or pre-retinal haemorrhage and/or rubeosis; NVD <1/4 DA + vitreous and/or pre-retinal haemorrhage and/or rubeosis;
* BCVA at baseline ≥ 24 Early Treatment Diabetic Retinopathy Study (ETDRS) letters score (approximate Snellen equivalent 20/320);
* Type I or Type II diabetic subjects of either gender;
* Age ≥ 18 years;
* Ability to provide written informed consent;
* Ability to return for all clinical trial visits;

Exclusion Criteria:

* Any intraocular surgery within 6 months before trial enrolment, including:

Prior scatter (panretinal) or focal/grid photocoagulation; Eyes who have received yttrium aluminum garnet (YAG) laser, or peripheral retinal cryoablation, or laser retinopexy (for retinal tears only);

* Fibrovascular proliferation with retinal traction;
* Other cause of retinal NV (retinal vein occlusion, radiation retinopathy or others);
* Atrophy/scarring/fibrosis/ hard exudates involving the centre of the macula;
* Significant media opacities or inadequate pupillary dilation, which might interfere with visual acuity, assessment of toxicity or fundus photography;
* Any likelihood that the subject will require cataract surgery within the following 1 year;
* Diabetic macular edema (DME) with central involvement, i.e., central macular thickness (Central Point Thickness) > 300 µm (Stratus OCT) equivalent values measured by spectral domain (SD)-OCT, adjusted according to the SD-OCT machine used;
* Previous vitrectomy;
* Intraocular pressure > 21 mmHg;
* Previous anti-VEGF therapy within the last 3 months;
* Known serious allergies or history of hypersensitivity to fluorescein used in angiography, or to components of Lucentis® formulation;
* Acute ocular or periocular infection;
* Previous filtering surgery (e.g., trabeculectomy) or placement of a glaucoma drainage device (e.g., tube-shunt surgery); General Exclusion Criteria
* Systolic BP > 170 mmHg or diastolic BP > 100 mmHg;
* HbA1C level >11% or recent signs of uncontrolled diabetes;
* Any of the following underlying systemic diseases:

History or evidence of severe cardiac disease, e.g. New York Heart Association (NYHA) Functional Class III or IV, clinical or medical history of unstable angina, acute coronary syndrome, myocardial infarction, or revascularization procedure within 6 months prior to baseline, or ventricular tachyarrhythmia requiring treatment; History or evidence of clinically significant peripheral vascular disease such as intermittent claudication or prior amputation; Renal failure requiring dialysis or renal transplant or renal insufficiency with creatinine levels > 2.0 mg/dl at screening; Stroke (within 12 months of trial entry); Any major surgical procedure within one month before trial enrolment;

* Subject with a condition (such as advanced, severe or unstable disease or its treatment) or is in a situation which may put him/her at significant risk, which may confound the study results or may interfere significantly with the subject's participation in the study;
* Previous radiation to the head in the region of the study eye;
* Use of any other investigational drugs within the last 3 months (for DR or other condition);
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases;
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Regression of neovascularization | 12-month treatment
  Defined as any decrease in the area of neovascularization

SECONDARY OUTCOMES:
Changes in Best Corrected Visual Acuity (BCVA) | 12-Month treatment
Time to complete neovascularization regression | 12-Month treatment
Recurrence of neovascularization | 12-Month treatment
Macular retinal thickness | 12-Month treatment
Need of treatment for Diabetic Macular Edema | 12-Month treatment
Need of vitrectomy due to the occurrence of vitreous hemorrhage, tractional retinal detachment or other complications of Diabetic Retinopathy. | 12-Month treatment
Adverse events related to the treatments | 12-Month treatment

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD, PhD, Study Chair — Association of Innovation and Biomedical Research on Light and Image
Locations (13):
- France (3):
  - Department of Ophthalmology, University Hospital, CHU Dijon, Dijon
  - Department of Ophthalmology, Lariboisière Hospital, Paris
  - Centre d'Investigation Clinique - Centre National d'Ophtalmologie des Quinze-Vingts, Paris
- Italy (3):
  - Department of Ophthalmology, University Vita Salute - Scientific Institute of San Raffael, Milan
  - Centre for Clinical Trials, Department of Ophthalmology, University of Padova, Padua
  - G.B.Bietti Eye Foundation - IRCCS, Rome
- Portugal (4):
  - Centre for Clinical Trials - Association for Innovation and Biomedical Research on Light and Image, Coimbra
  - Espaço Médico de Coimbra, Coimbra
  - Instituto de Retina de Lisboa, Lisbon
  - Serviço de Oftalmologia,Hospital de Vila Franca de Xira, Vila Franca de Xira
- United Kingdom (3):
  - Ophthalmology Clinical Trials Unit Frimley Park Hospital Foundation Trust, Frimley
  - Clinical Trial Unit, Dep. Ophth., Gloucestershire Hospitals NHS Foundation Trust, Gloucestershire
  - Laser and Retinal Research Unit, King's Health Partners, London